CLINICAL TRIAL: NCT07161908
Title: Early Detection and Prevention of Health Complications in Preterm Infants - Controlled Remote Monitoring and Optimization of Oxygen Therapy
Brief Title: Controlled Remote Monitoring and Optimization of Oxygen Therapy in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: České Budějovice Hospital (Other); University Hospital Olomouc (Other); Institute for the Care of Mother and Child, Prague, Czech Republic (Other); General University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UZIS 2025/1
Record Dates: First submitted 2025-08-12; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: BPD - Bronchopulmonary Dysplasia; Pulmonary Hypertension
Keywords: BPD; Bronchopulmonary Dysplasia; preterm infants; oxygen therapy; telemedicine; remote monitoring; pulmonary hypertension; Czech Republic
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Controlled remote oxygen therapy (Experimental): The patients will be following study protocol of optimization of oxygen therapy.
  Interventions: Device: Pulse oximeter

INTERVENTIONS:
Device: Pulse oximeter — To ensure proper treatment, the infant will be continuously monitored with a pulse oximeter. Based on oxygen saturation levels, the treatment may be adjusted according to pre-established protocols. It is required that the saturation stays above a certain value for more than 95 % of the 12-hour measurement period. If the defined saturation values are reached, the parents will reduce the oxygen flow by one degree for 20 minutes in the hospital/home setting (20 minute test) and if the saturation values remain at 93 % or more during this period, overnight 12 hour monitoring will also be performed to confirm stable saturation values of 93 % or more for 95 % or more of the monitoring time.
  Thanks to modern specialized pulse oximeters, it is possible to ensure accurate, long-term, remotely managed monitoring of the infant and to interactively optimize oxygen therapy based on current oxygen saturation levels.

SUMMARY:
The project is a national, prospective, multicenter, interventional pilot project focused on controlled remote monitoring and optimization of oxygen therapy for premature infants in the Czech Republic. The primary aim of the project is to prepare, test, and develop a proposal for a national methodology for the care of preterm newborns. This will reduce health risks in premature infants and minimize the negative impacts on the overall development of the child and the family of the premature infant.

DETAILED DESCRIPTION:
The project is a national, prospective, multicenter, interventional pilot project focused on remote monitoring and optimization of oxygen therapy for premature infants in the Czech Republic.

The main goal of the project is validation of the possibility and organization of remotely managed home oxygen therapy and its optimization, aiming for its earlier termination.

The project will be running in 4 perinatology centers in the Czech Republic. It is expected that 70 premature infants diagnosed with bronchopulmonary dysplasia will participate. The infant must transition to low-flow nasal cannulas to be discharged to home care. Oxygen therapy will be adjusted based on pre-established protocols aiming for earlier and safer termination of oxygen therapy through precise remote continual monitoring.

The project is supported by the European Social Fund (Operational Program Employment Plus) and the state budget of the Czech Republic and is registered by the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.02.02/00/22_005/0002020.

The study has been reviewed and approved by multiple local ethical committees. The listed IRB represents the lead national ethical committee overseeing the trial.

ELIGIBILITY:
Inclusion Criteria:

* infants born before 31+6 weeks gestation
* signed consent for participation in the project and consent for the processing of personal data
* diagnosed with bronchopulmonary dysplasia
* type of pulmonary ventilation - low-flow nasal cannulas

Exclusion Criteria:

* unsigned consent for participation in the project and/or consent for the processing of personal data
* child diagnosed with conditions other than bronchopulmonary dysplasia (BPD) at high risk of long-term hypoxia - selected chronic cardiovascular, neurological, and muscular diseases, e.g., significant congenital heart defects, congenital central nervous system developmental disorders, genetic diseases associated with the risk of hypoventilation, central apneas, severe early obstructive sleep apnea
* other chronic respiratory diseases besides BPD - e.g., cystic fibrosis, chronic aspiration
* insufficient therapy through long-term home oxygen therapy
* tracheostomy

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Average duration of controlled oxygen therapy in a premature infant | From the enrollment to 4 weeks after discontinuation of home oxygen therapy application in child (complete weaning from oxygen supply)
  Number of days a premature infant stays on oxygen therapy

SECONDARY OUTCOMES:
Average number of failures in premature infants before the termination of controlled oxygen therapy | From the enrollment to 4 weeks after discontinuation of home oxygen therapy application in child (complete weaning from oxygen supply)
  Failure is defined as the need to return to the original flow rate before the last reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Plavka, prof., Study Director — General Hospital University in Prague; Jana Tuková, Ph.D., Study Chair — General Hospital University in Prague
Locations (4):
- Czechia (4):
  - České Budějovice Hospital, České Budějovice, Czech Republic
  - University Hospital Olomouc, Olomouc, Czech Republic
  - General University Hospital, Prague, Czech Republic
  - Institute for the Care of Mother and Child, Prague, Czech Republic